CLINICAL TRIAL: NCT00974662
Title: Evaluation of the Safety and Efficacy of WST11-mediated Vascular Targeted Photodynamic Therapy on Obstructing Endobronchial Non-Small Cell Lung Cancer
Brief Title: Study Using WST11 in Patients With Obstructing Endobronchial Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early end of enrolment with regards to difficulty met to enrol patients.
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN903 LCM201
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Lung Cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — padeliporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WST11 (Experimental): Treatment with WST11-mediated VTP
  Interventions: Drug: WST11

INTERVENTIONS:
Drug: WST11 — WST11-mediated VTP will consists of the combination of a single IV administration of WST11 at doses of 5, 7.5 & 10 mg/kg, using 753 nm laser light at a fixed power of 250 mW/cm and escalating fixed energy dose (200 Joules/cm and 300 Joules/cm) locally delivered to the obstructing tumor through an optical fiber placed, during endoscopy, in the endoscope operating channel with visual control, possibly video-transmission assisted. The fiber illuminating diffusion length is fixed (2 cm).
  Other Names: WST11-mediated VTP

SUMMARY:
The aim of this study is to determine the dose of WST11 and light energy necessary to obtain desobstruction of the bronchial lumen using Vascular Targeted Photodynamic therapy in obstructive Non-Small Cell Lung Cancer.

DETAILED DESCRIPTION:
This study is designed as a multicentre, exploratory phase IIa, open label, single intravenous (IV) dose, escalating treatment regimen (Treatment regimen = a single dose of WST11 associated with a particular laser light energy) with a one month follow-up.

Six escalating treatment regimens will be followed: 3 WST11 doses (5 mg/kg; 7.5 mg/kg and 10 mg/kg) combined with 2 light energies (200 Joules/cm and 300 Joules/cm)

The patient will be treated under local anesthesia. The light is produced using a specific laser at a wavelength of 753 nm at a fixed power of 250 mW/cm and locally delivered to the obstructing tumor through an optical fiber placed, during endoscopy, in the endoscope operating channel with visual control, possibly video-transmission assisted. The fiber illuminating diffusion length is fixed (2 cm).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven lung cancer
* Inoperable
* Non-Small Cell Cancer
* Partial or total bronchial obstruction responsible for functional signs
* T1 to T4, N0-N3, M0-M1
* Patients with functional signs: hemoptysis, infection, cough and, above all, dyspnea
* Contralateral metastases not representing a contraindication insofar as they do not represent a risk of impairment of respiratory function during treatment
* The Karnofsky index should be greater than or equal to 40
* Patients should agree to and tolerate repeated bronchial endoscopy (a disadvantage of all endoscopic treatments)
* Male or female patients aged over 18 years, female patients should not be pregnant (menopause or contraception)
* Patients should have given their written consent to take part in the study

Exclusion Criteria:

* Tracheal lesions and lesions affecting the carina tracheae
* Patients with painful bone metastases (not an absolute criterion since the extent of dyspnea is the decisive element)
* Patients with brain metastases
* Patients having undergone pneumonectomy
* Patients undergoing chemotherapy or radiotherapy or having undergone chemotherapy less than 4 weeks before the procedure or radiotherapy less than 4 weeks before the procedure
* Patients with risk of large vessel erosion or perforation resulting from lesion topography
* In case of allergy to the photosensitizer
* Leukopenia (WBC<2000), Thrombocytopenia (< 100 000), PT > 1.5 normal, Fibrinogen < 2g/l, a PTT > 1.5 ULN (Upper Limit of Normal)
* Renal insufficiency
* Hepatic insufficiency
* Patients having already received 70 Gy on the lesion
* Existing tracheoesophageal or bronchoesophageal fistula
* Emergency treatment of patients with severe acute respiratory distress caused by an obstructing endobronchial lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The percentage of bronchial obstruction before and after treatment represents the main evaluation parameter. | Week 1, Month 1

SECONDARY OUTCOMES:
The evaluation of safety will be based on adverse events reporting throughout the duration of the study, on the monitoring of vital signs and ECGs, on laboratory tests,clinical examination and chest X Ray. | Screening-Month 3
Quality of life will be assessed through the validated patient questionnaires | Baseline, Week 1, Month 1 & Month 3
To assess pharmacokinetic parameters of WST11 | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Michel Leroy, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France